CLINICAL TRIAL: NCT07050082
Title: Cystoinflation to Prevent Bladder Injury in Cases of Placenta Accreta Spectrum , a Randomized Controlled Trial
Brief Title: Cystoinflation to Prevent Bladder Injury in Cases of Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Sharawy Abdelrahman, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cystoinflation in PAS cases
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2023-06

CONDITIONS: Bladder Injury; Accreta, Placenta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder filling (Experimental): 42 case of PAS , bladder dissection done after filling bladder with 200 cc saline
  Interventions: Procedure: Bladder dissection after filling with 200 cc saline solution
- Non bladder filling (Active Comparator): 42 case of PAS , bladder dissection done with empty bladder
  Interventions: Other: Bladder dissection with empty bladder

INTERVENTIONS:
Procedure: Bladder dissection after filling with 200 cc saline solution — Bladder filling after entering peritoneal cavity, then bladder dissection done to avoid bladder injury
  Other Names: Bladder filling; Cystoinflation; Bladder dissection
  Arms: Bladder filling
Other: Bladder dissection with empty bladder — After entering peritoneal cavity, bladder dissection done with empty bladder
  Other Names: Classic bladder dissection
  Arms: Non bladder filling

SUMMARY:
Placenta accreta spectrum (PAS) disorders are associated with a high risk of bladder injury .leading to increased morbidity. Cystoinflation, involving controlled retrograde bladder filling, has been proposed as a technique to improve intraoperative visualization and reduce bladder injuries.

Objective To evaluate the efficacy and safety of cystoinflation in preventing bladder injuries in cases of PAS.

Methods This randomized controlled trial included 84 women diagnosed with PAS, allocated equally into cystoinflation and control groups. The cystoinflation group underwent bladder filling with 200 mL saline to facilitate dissection, while the control group did not. Primary outcome measures included the incidence of bladder injury, operative time. Data were analyzed using appropriate statistical tests with significance set at p<0.05.

DETAILED DESCRIPTION:
The global incidence of placenta accreta spectrum (PAS) disorders are rising in parallel with the increasing rates of cesarean delivery, posing significant challenges in obstetric practice due to its association with severe maternal morbidity and mortality . PAS encompasses a spectrum of abnormal placental adherence, which can lead to life-threatening hemorrhage during delivery.

In response to the limitations of traditional terminology (placenta accreta, increta, percreta), the International Federation of Gynecology and Obstetrics introduced a standardized classification under the umbrella of PAS disorders, aiming to improve diagnostic clarity and clinical management.

Surgical management recognized as the standard of care for invasive placentation .However, this procedure carries a substantial risk, with severe maternal morbidity rates reaching 40-50%, primarily due to hemorrhage and injury to adjacent organs. In extreme cases, maternal mortality may reach up to 7% .The complexity of the surgery is heightened by the high risk of adjacent organ injury, with an adjusted odds ratio of 8.2 for damage to nearby structures .

Among these complications, urinary tract injury is notably prevalent. Risk factors include the depth and lateral extension of placental invasion, the extent of intraoperative blood loss, and the number of prior cesarean sections . Urinary tract trauma occurs in approximately 29% of PAS-related surgeries, with bladder lacerations accounting for 76%, ureteral injuries for 17%, and genitourinary fistulas for 5% . Although injuries to the bowel, pelvic vasculature, and nerves are less common, they remain clinically significant .

Bladder injury, in particular, has profound implications, contributing to prolonged operative time, urinary tract infections, voiding dysfunction, and extended catheterization, all of which adversely affect a patient's physical and psychological well-being .While routine preoperative bladder catheterization aids in visualizing the surgical field, it often fails to prevent bladder injury in cases with dense adhesions.

This study aims to assess the efficacy and safety of bladder filling with 200 cc saline during bladder dissection in women diagnosed with PAS.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 34 weeks or more
* BMI 18.5-29.9
* Placcenta accreta diagnosed by ultrasound
* Previous caesarian section
* General anaesthetia

Exclusion Criteria:

* medical disorders
* History of bladder injury or previous bladder surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of bladder injury in two groups | 18 months
  Comparing incidence of bladder injury in cases of PAS with and without bladder filling

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided